CLINICAL TRIAL: NCT03804372
Title: Prospective Study on the Incidence of Hepatitis B Virus Reactivation in Untreated Patients With Diffuse Large B-Cell Lymphoma/Chronic Lymphoid Leukemia HBsAg-positive Treated With Rituximab, Chemotherapy and Tenofovir Alafenamide
Brief Title: The Incidence of Hepatitis B in Diffuse Large B-Cell Lymphoma/Chronic Lymphoid Leukemia HBsAg-positive Treated With Rituximab, Chemotherapy and Tenofovir Alafenamide
Acronym: CLL1818
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low enrollment rate
Sponsor: Gruppo Italiano Malattie EMatologiche dell'Adulto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLL1818
Record Dates: First submitted 2019-01-08; First posted 2019-01-15 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Large-B-cell Diffuse Lymphoma; Chronic Lymphoid Leukemia
Keywords: diffuse Large B-Cell Lymphoma; chronic Lymphoid Leukemia HBsAg-positive; Rituximab; chemotherapy; alafenamide; hepatitis B virus reactivation
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse; Leukemia, B-Cell | interventions — Rituximab; Drug Therapy; tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study group (Experimental): Patients will receive Rituximab+Chemotherapy+TAF for 6 months, followed by TAF as monotherapy for further 12 months. All subjects will receive TAF 1-3 weeks before Rituximab+Chemotherapy and withdrawn 12 months after the completion of chemotherapy.
  Interventions: Drug: Rituximab; Drug: Chemotherapy; Drug: Tenofovir alafenamide

INTERVENTIONS:
Drug: Rituximab — Patients will receive Rituximab+Chemotherapy+TAF for 6 months, followed by TAF as monotherapy for further 12 months. All subjects will receive TAF 1-3 weeks before Rituximab+Chemotherapy and withdrawn 12 months after the completion of chemotherapy.
Drug: Chemotherapy — Patients will receive Rituximab+Chemotherapy+TAF for 6 months, followed by TAF as monotherapy for further 12 months. All subjects will receive TAF 1-3 weeks before Rituximab+Chemotherapy and withdrawn 12 months after the completion of chemotherapy.
Drug: Tenofovir alafenamide — Patients will receive Rituximab+Chemotherapy+TAF for 6 months, followed by TAF as monotherapy for further 12 months. All subjects will receive TAF 1-3 weeks before Rituximab+Chemotherapy and withdrawn 12 months after the completion of chemotherapy.

SUMMARY:
In this study, we will evaluate the incidence of hepatitis B virus reactivation within the first 6 months of treatment with rituximab, standard chemotherapy and TAF in patients with diffuse Large B-Cell Lymphoma/Chronic Lymphoid Leukemia HBsAg-positive.

DETAILED DESCRIPTION:
This is a prospective, multicenter, interventional, single arm, evaluating the incidence of hepatitis B virus (HBV) reactivation within the first 6 months treatment period in HBsAg positive patients treated for DLBCL/Chronic Lymphoid Leukemia with Rituximab, standard chemotherapy, and TAF.

Approximate duration of the recruitment period based on the number of patients available The duration of the recruitment period has been estimated at 12 months.

Patients will receive Rituximab+Chemotherapy+TAF for 6 months, followed by TAF as monotherapy for further 12 months. All subjects will receive TAF 1-3 weeks before Rituximab+Chemotherapy and withdrawn 12 months after the completion of chemotherapy. Then patients will be also observed for further12 months

ELIGIBILITY:
Inclusion Criteria:

* Signed written informed consent according to ICH/EU/GCP and national local laws.
* Male/non-pregnant/non-lactating female subjects >18 years old with newly diagnosed DLBCL/Chronic Lymphoid Leukemia who are going to receive treatment with rituximab in combination with chemotherapy.
* HBsAg positivity, serum HBV-DNA negative or positive (<2000/IU), and normal liver function, including alanine aminotransferase(ALT), aspartate aminotransferase(AST) and bilirubin. (inactive carriers).
* No previous treatment with antiviral drugs for HBV infection.
* Patients with satisfactory renal function.

Exclusion Criteria:

* Hepatic insufficiency for any reason
* History of other liver diseases such as hepatitis C, D, autoimmune hepatitis, primary biliary cirrhosis, Wilsons' disease
* Positive viral markers, such as IgM antibody to hepatitis A virus, hepatitis C virus, IgG antibody to hepatitis D virus, IgM antibody to hepatitis E virus, or antibody to HIV
* Pregnant or breastfeeding women
* Other major systemic diseases, such as active infection, significant cardiac disease, neurological deficit or psychiatric disorder, that the investigators consider being a significant risk
* Patients with moderate or severe renal failure.
* Intolerance to any of the components of the therapeutic regimen. Treatment with any investigational medicinal product (unapproved) in the last 30 days.
* Any other disorder that, in the investigator's opinion, makes the patient ineligible for recruitment or that could interfere in his/her participation or in the conclusion of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2020-07-07 (Actual); Primary Completion 2024-05-22 (Actual); Study Completion 2024-05-22 (Actual)

PRIMARY OUTCOMES:
Percentage of patients presenting hepatitis B virus reactivation | Within 6 months following the start of treatment
  Assessment of the percentage of patients presenting HBV reactivation within 6 months following the start of treatment with Rituximab, chemotherapy and TAF in in DLBCL and Chronic Lymphoid Leukemia patients.

SECONDARY OUTCOMES:
Percentage of patients presenting hepatitis B virus reactivation | After 12 months following the study entry and start of treatment
  Assessment of the percentage of patients presenting HBV reactivation during and after the 12-month treatment of TAF as a single agent in in DLBCL and Chronic Lymphoid Leukemia patients
Number of patients stratified by DLBCL and Chronic Lymphoid Leukemia with hepatitis related to the HBV infection or with liver failure during their participation in the study. | After 31 months from study entry
Percentage of patients in which chemotherapy is delayed due to HBV-reactivation. | After 31 months from study entry
  In terms of percentage of patients with a delay of at least 7 days between chemotherapy cycles stratified by DLBCL and chronic lymphoid leukemia.
Number of patients with DLBCL and with Chronic Lymphoid Leukemia who survive | After 31 months from study entry
Number of patients experiencing adverse events. | After 31 months from study entry

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Gentile, Study Chair — Università Sapienza di Roma; Alessandra Micozzi, Study Director — Università Sapienza di Roma
Locations (31):
- Italy (31):
  - Aon Ss. Antonio E Biagio E C. Arrigo - Alessandria - Soc Ematologia, Alessandria
  - Aou Ospedali Riuniti "Umberto I - G.M. Lancisi - G. Salesi"- Ancona - Sod Clinica Ematologica, Ancona
  - Area Vasta N. 5 Ascoli Piceno - S. Benedetto Del Tronto, Presidio Ospedaliero Av5 Osp. Gen. Prov.Le "C.G.Mazzoni" - Uoc Ematologia, Ascoli Piceno
  - Irccs Centro Di Riferimento Oncologico Di Aviano - Sosd Oncoematologia Trapianti Emopoietici E Terapie Cellulari, Aviano
  - Aou Consorziale Policlinico - Bari - Uo Ematologia Con Trapianto, Bari
  - Irccs Oncologico Istituto Tumori Giovanni Paolo Ii - Bari - Uo Ematologia, Bari
  - Asl Brindisi, Ospedale 'Perrino' - Brindisi - Uo Ematologia, Brindisi
  - Ctc U.O Di Ematologia Con Trapianto Di Midollo Osseo - Catania, Catania
  - Aou Arcispedale Sant'Anna - Cona (Fe) - Uoc Ematologia E Fisiopatologia Della Coagulazione, Cona
  - Aou Ospedali Riuniti - Foggia - Uoc Ematologia, Foggia
  - Asl Lecce, Ospedale 'V. Fazzi' - Uo Ematologia, Lecce
  - Ao Ospedali Riuniti "Papardo Piemonte" - Po Papardo - Messina - Sc Ematologia, Messina
  - Ao Di Rilievo Nazionale Antonio Cardarelli - Napoli - Uoc Ematologia Con Trapianto Di Midollo, Napoli
  - Aou Federico Ii - Napoli - Uoc Ematologia, Napoli
  - Aou Maggiore Della Carita' Di Novara - Scdu Ematologia, Novara
  - Asl Salerno, Presidio Ospedaliero Tortora Pagani - Ematologia, Pagani
  - Ao Ospedali Riuniti Villa Sofia Cervello - Palermo - Uo Ematologia Con Utmo, Palermo
  - Fondazione Ircss Policlinico San Matteo - Pavia - Uo Ematologia, Pavia
  - Asl Pescara, Presidio Ospedaliero 'Spirito Santo' - Uoc Ematologia Clinica, Pescara
  - Ausl Di Reggio Emilia - Arcispedale Santa Maria Nuova, Irccs - Sc Ematologia, Reggio Emilia
  - Ausl Della Romagna, Ospedale "Infermi" - Rimini - Uo Ematologia, Rimini
  - Ao San Camillo Forlanini - Roma - Uoc Ematologia E Trapianto Cellule Staminali, Roma
  - Aou Policlinico Tor Vergata - Roma - Uoc Trapianto Cellule Staminali, Roma
  - Aou Sant'Andrea - Roma - Uoc Ematologia, Roma
  - Asl Roma 2, Ospedale S. Eugenio- Ospedale S.Eugenio - Uoc Ematologia, Roma
  - Fondazione Policlinico Universitario Agostino Gemelli Irccs - Roma - Area Ematologica, Roma
  - Università degli Studi "Sapienza" - Dip Biotecnologie Cellulari ed Ematologia - Divisione di Ematologia, Roma
  - Ente Ecclesiastico Casa Sollievo Della Sofferenza - San Giovanni Rotondo - Ematologia, San Giovanni Rotondo
  - Aou Città Della Salute E Della Scienza, Ospedale S. Giovanni Battista Molinette - Torino - Sc Ematologia - Università Degli Studi Di Torino, Torino
  - Aou Integrata Di Verona, Policlinico G.B. Rossi - Uoc Ematologia, Verona
  - Aulss 8 Berica - Ospedale Di Vicenza - Uoc Ematologia, Vicenza

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Picardi M, Giordano C, Della Pepa R, Pugliese N, Leone A, Delle Cave G, Iula R, Pane F, Gentile G. Regarding "Hepatitis B Surface Antigen Positivity Is an Independent Unfavorable Prognostic Factor in Diffuse Large B-Cell Lymphoma in the Rituximab Era". Oncologist. 2021 Jun;26(6):e1083-e1084. doi: 10.1002/onco.13710. Epub 2021 Feb 24. PMID 33559286